CLINICAL TRIAL: NCT05391139
Title: Acute Effects of Dual Task During Upper Limb Strengthening on Physical Function and Pain in Patients With Elbow Joint Fracture
Brief Title: Acute Effects of Dual Task on Physical Function in Patients With Elbow Joint Fracture
Acronym: ACEDTELBOW
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Laura López-Bueno, Principal Investigator, University of Valencia
Other Study IDs: ID0002
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Elbow Fracture
MeSH Terms: conditions — Elbow Fractures

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Elbow injuries account for up to 15% of emergency consultations. The complexity of this joint and the subtle imaging findings present even in severe injuries make diagnosis difficult and can delay treatment, causing pain and functional impotence. Appropriate deterioration mitigation strategies include, but are not limited to, strengthening programs of sufficient intensity to stimulate anabolism and limit muscle loss and increase strength. The general recommendation for increasing muscle strength and neural adaptations in healthy subjects after sustaining an elbow fracture is moderate to heavy load resistance training with loads approximating 60%-80% of the one repetition maximum ( 1RM). However, high joint stress would be challenging and increase the risk of adverse consequences in such patients, so strategies are still needed to meet the challenges of effectively and safely adapting training loads to safely enable improvement. without requiring high joint stress. Resistance band work, coupled with the use of dual tasks, is a novel approach used during resistance training, especially among healthy populations, with promising results. The purpose of the study is to evaluate acute neuromuscular responses, pain intensity and RPE in patients with elbow joint fracture, with or without surgical approach, with different strategies to strengthen the upper limb.

Candidates for this study will be men and women over 18 years of age who have been diagnosed with a fracture of the elbow joint (types 1-3 and types 2-1 according to Müller's OA fracture classification), with or without a surgical approach and with date of injury and completion of their physiotherapy program in 2022-2023, and who begin their physiotherapy treatment between weeks 7 to 9 post-fracture.

DETAILED DESCRIPTION:
Elbow injuries account for up to 15% of emergency consultations. The complexity of this joint and the subtle imaging findings present even in severe injuries make diagnosis difficult and can delay treatment, causing pain and functional impotence. Appropriate deterioration mitigation strategies include, but are not limited to, strengthening programs of sufficient intensity to stimulate anabolism and limit muscle loss and increase strength. The general recommendation for increasing muscle strength and neural adaptations in healthy subjects after sustaining an elbow fracture is moderate to heavy load resistance training with loads approximating 60%-80% of the one repetition maximum (1RM). However, high joint stress would be challenging and increase the risk of adverse consequences in such patients, so strategies are still needed to meet the challenges of effectively and safely adapting training loads to safely enable improvement. without requiring high joint stress. Resistance band work, coupled with the use of dual tasks, is a novel approach used during resistance training, especially among healthy populations, with promising results. The purpose of the study is to evaluate acute neuromuscular responses, pain intensity and RPE in patients with elbow joint fracture, with or without surgical approach, with different strategies to strengthen the upper limb.

Candidates for this study will be men and women over 18 years of age who have been diagnosed with a fracture of the elbow joint (types 1-3 and types 2-1 according to Müller's OA fracture classification), with or without a surgical approach and with date of injury and completion of their physiotherapy program in 2022-2023, and who begin their physiotherapy treatment between weeks 7 to 9 post-fracture. The patients will voluntarily participate in the study, which will be carried out at the Hospital Clínico Universitario de Valencia, during the months of May 2022 to May 2023. All participants will be informed about the objectives and content of the research and information will be obtained. written informed consent. The study will conform to the Declaration of Helsinki and will be approved by the local ethics committee. Participants will be excluded if they have any involvement in the contralateral upper limb, if they have already had/have any other injury to the elbow or other anatomical part of the affected MS (in the last year), and if they have any other condition or disease in the which there is a contraindication to physical exercise.

Also if they participate in physiotherapy programs external to the one carried out by us or in other research studies. In addition, if there is evidence of a severe failure in bone consolidation (separation greater than 5 mm), if there is neural injury, CRPS (Complex Regional Pain Syndrome), severe open fracture with muscle and periosteal loss, clinical picture not competent for physiotherapy by diagnosis doubtful and severe congenital instability of MMSS. The study consists of observational session will be held. The experimental protocol begins with the evaluation of neuromuscular responses, self-perceived pain intensity and RPE from the use of different intensities of elastic resistance, during elbow flexion and extension, at a controlled speed of 1.5 sec/phase. For this purpose, 1.5 m long elastic bands will be available, which will be previously stretched to approximately 25% of their initial length. This intensity is selected because it appears to correspond to the appropriate weight which is equivalent to 30% of 1RM and is considered a light intensity. At the end of each set of the exercise, you will be asked about RPE (Borg CR10) and pain in the joint. The exercises must be performed with the available range of movement of the subject. Participants are asked to move their body and trunk as little as possible and to perform the exercise smoothly, without stopping or accelerating. Elbow flexion will be performed in a sitting position and extension in the supine position, both stable positions, with exact fastening of the bands on the panel of the Rocher Cage, located in the therapeutic room.

The subjects, in a counterbalanced way, will perform 4 different conditions, with 10 minutes of rest between them: the possibilities are 1) perform all possible repetitions of elbow flexion with the appropriate band; 2) perform all possible repetitions of elbow flexion with the appropriate band, and following a dual task; 3) perform as many elbow extension reps as possible with the appropriate band; 4) perform as many elbow extension repetitions as possible with the appropriate band, and following a dual task.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for this study will be men and women over 18 years of age who have been diagnosed with a fracture of the elbow joint. The patients will voluntarily participate in the study, which will be carried out at the Hospital Clínico Universitario de Valencia, during the months of May 2022 to May 2023. All participants will be informed about the objectives and content of the research and information will be obtained. written informed consent. The study will conform to the Declaration of Helsinki and will be approved by the local ethics committee.

Exclusion Criteria:

* Participants will be excluded if they have any involvement in the contralateral upper limb, if they have already had/have any other injury to the elbow or other anatomical part of the affected MS (in the last year), and if they have any other condition or disease in the which there is a contraindication to physical exercise. Also if they participate in physiotherapy programs external to the one carried out by us or in other research studies. In addition, if there is evidence of a severe failure in bone consolidation (separation greater than 5 mm), if there is neural injury, CRPS (Complex Regional Pain Syndrome), severe open fracture with muscle and periosteal loss, clinical picture not competent for physiotherapy by diagnosis doubtful and severe congenital instability of upper members.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidates for this study will be men and women over 18 years of age who have been diagnosed with a fracture of the elbow joint (types 1-3 and types 2-1 according to Müller's OA fracture classification), with or without a surgical approach and with date of injury and completion of their physiotherapy program in 2022-2023, and who begin their physiotherapy treatment between weeks 7 to 9 post-fracture.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Mobility | 1 day
  The experimental protocol begins with the evaluation of neuromuscular responses, self-perceived pain intensity and RPE from the use of different intensities of elastic resistance, during elbow flexion and extension. This intensity is selected because it appears to correspond to the appropriate weight which is equivalent to 30% of 1RM and is considered a light intensity.

SECONDARY OUTCOMES:
Kinesiophobia | 1 day
  Kinesiophobia will be evaluated mainly through the Spanish version of the Kinesiophobia Tampa Scale in a selfrecorded manner. This instrument has shown adequate reliability (showing an internal consistency of α=0.79). The total score ranges between 11 and 44 points, with higher levels of kinesiophobia the higher the score obtained on the scale. In addition, kinesiophobia specific to the type of exercise performed will be assessed, with a self-perceived scale from 0 to 10, where patients will indicate the fear of performing all possible repetitions during a strength exercise.
Shoulder functionality | 1 day
  It will be evaluated using the DASH questionnaire in Spanish. The assessment of the ability to perform various tasks (open a new or very tight jar, write, turn a key, prepare food, etc.), The score can range between 30 and 150 points.
  A higher score indicates a higher level of disability and severity, while a lower percentage indicates a low level of disability. This questionnaire has shown adequate reliability (showing an internal consistency of α=0.96).
Self-reported pain intensity | 1 day
  The patient marks a point on the scale and subsequently, the clinician or researcher quantifies the number of mm indicated by the patient.Therefore, the self-perceived pain intensity range travels from 0-100 mm. VAS is the most widely used so far in research to assess pain intensity.
Measurement of range of motion | 1 day
  The degrees of movement (ROM) of the following joints shall be actively and passively measured by means of a manual goniometer: elbow (flexion and extension), forearm (pronation and supination), wrist (flexion and extension), metacarpophalangeal (flexion), proximal intephalangeal (flexion) and distal interphalangeal (flexion).
Isometric elbow extension/flexion force | 1 day
  They will be evaluated with a portable handheld dynamometer. The tests will be carried out against a fixed resistance:
  the participants were with their elbows at 90º, in a sitting position with an upright posture, without a backrest and with both feet placed flat on the floor, with force exerted against a fixed table. 3 maximum contractions of 5 seconds will be performed, separated by 1 minute of rest, selecting the average value of these 3 for later analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Laura López-Bueno, Principal Investigator — University of Valencia
Locations (1):
- Laura López-Bueno, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No